CLINICAL TRIAL: NCT05682027
Title: Ultrasound as Diagnostic Tool in Diaphragm Dysfunction: a Prospective Observational Study.
Brief Title: Ultrasound as Diagnostic Tool in Diaphragm Dysfunction
Acronym: ULTRASONIC
Status: Completed | Type: Observational
Sponsor: Isala (Other)
Responsible Party: Principal Investigator, Wytze de Boer, M.D., Isala
Other Study IDs: Diaphragm 001
Record Dates: First submitted 2022-12-27; First posted 2023-01-12 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Diaphragm Disease
Keywords: diaphragm dysfunction; ultrasound; fluoroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients suspected of diaphragm dysfunction: After inclusion, participants will be evaluated for diaphragm dysfunction with fluoroscopy, as in standard of care. Additionally, during the same hospital visit ultrasound will be performed.
  The sonographer and the radiologist assessing the ultrasound and fluoroscopy, respectively, will be blinded to each other's' test results. Further assessment, and possible treatment, for diaphragm dysfunction is performed at the discretion of the treating physician.
  The primary outcome is the concordance of diaphragm paralysis as determined by ultrasound compared with the construct for diaphragm paralysis based on traditional measurements.
  Interventions: Diagnostic Test: ultrasound of the diaphragm

INTERVENTIONS:
Diagnostic Test: ultrasound of the diaphragm — Parameters measured during ultrasound:
  Thickening fraction; End-expiratory thickness, and; Diaphragm excursion.

SUMMARY:
The diaphragm is the main muscle for inspiration and vital for ventilation. Multiple diagnostic modalities can be performed in the work-up of suspected diaphragm dysfunction. Fluoroscopy has traditionally been the method of choice in diagnosing diaphragm paralysis and is still widely used in clinical practice, while alternative non-invasive and accessible methods have been available. Superiority of ultrasound over fluoroscopy for the diagnosis of diaphragm dysfunction has been suggested.

The primary objective of this study is to investigate the construct validity of ultrasound in diaphragm paralysis.

DETAILED DESCRIPTION:
To study the sensitivity of ultrasound in diaphragm dysfunction we propose a prospective, operator-blinded, two-center, observational study. Participants will be evaluated for diaphragm dysfunction with fluoroscopy and pulmonary function testing as in standard of care. Additionally, ultrasound will be performed.

Construct validity The primary objective of this study is to investigate the construct validity of ultrasound in diaphragm paralysis. Validity is defined as the degree to which an instrument truly measure the construct(s) it purports to measure. In general, three different types of validity can be distinguished: content validity, criterion validity, and construct validity. Since evaluation with gold standard testing is invasive, as explained in the introduction, criterion validity testing not a feasible option. Therefore, in this study, we use construct validity to provide evidence of validity. Construct validity is defined as the degree to which the scores of an instrument (here: ultrasound) are consistent with scores of other instruments (here: pulmonary function tests, fluoroscopy). Construct validation is often considered less powerful, however, with strong theories and specific and challenging hypothesis, it is possible to acquire substantial evidence. Therefore, specific definitions of 'diaphragm paresis' and 'diaphragm paralysis' regarding diagnostic modalities are established in this protocol before the start of the study

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Suspicion of diaphragm dysfunction based on medical history and/or physical examination; as determined by the treating physician.

Exclusion Criteria:

* Inability for fluoroscopy (e.g. severely limited mobility, or unable to follow vocal instructions).
* Inability for diaphragm imaging (e.g. mechanical ventilation, or unable to follow vocal instructions).
* Those not able or unwilling to give written informed consent.
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our population consists of 18-years or older patients suspected of diaphragm dysfunction based on medical history and/or physical examination; as determined by the treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-21 (Actual)

PRIMARY OUTCOMES:
Concordance of diaphragm paralysis as determined by ultrasound compared with the construct for diaphragm paralysis based on traditional measurements | From referall till completion of diagnostic tests.
  Parameters:
  * Paralysis (ultrasound): Qualitative (visual): Paradoxal movement OR Quantitative: Diaphragm Excursion(DE) < 0cm (negative).
  * Paralysis (reference): (Physical examination suggestive of diaphragm dysfunction (i.e. paradoxal abdominal movement) OR Decrease in vital capacity of >15% when suspine) AND Paradoxal movement during fluoroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: wytze de Boer, M.D., Study Director — Isala
Locations (2):
- Netherlands (2):
  - Isala Klinieken, Zwolle, Overijssel
  - UCMG, Groningen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] de Boer WS, Parlevliet KL, Kooistra LA, Koster D, Nieuwenhuis JA, Edens MA, van den Berg JWK, Boomsma MF, Stigt JA, Slebos DJ, Duiverman ML. Ultrasound as diagnostic tool in diaphragm dysfunction: a prospective construct validity study. Respir Med. 2025 May;241:108083. doi: 10.1016/j.rmed.2025.108083. Epub 2025 Apr 4. PMID 40187575